CLINICAL TRIAL: NCT04797455
Title: Pilot Intervention for Parents of Psychiatrically-Hospitalized Youth
Brief Title: Parent Intervention for Psychiatrically-Hospitalized Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michele Berk, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59389
Record Dates: First submitted 2021-03-07; First posted 2021-03-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Adolescent - Emotional Problem; Suicide and Self-harm; Parenting
Keywords: suicide; Self-Injurious Behavior; Behavioral Symptoms
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Behavioral Symptoms | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PI+ Inpatient Treatment as Usual (Experimental): Standard inpatient treatment delivered in the context of an adolescent psychaitric inpatient unit plus an 4 session DBT-based parenting intervention PI)
  Intervention: Behavioral: DBT-Based Parenting Intervention
  Interventions: Behavioral: DBT-Based Parenting Intervention; Behavioral: Treatment as usual
- Inpatient Treatment alone (Active Comparator): No parenting intervention provided beyond what is part of the inpatient treatment as usual.
  Intervention: Behavioral: Treatment as Usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: DBT-Based Parenting Intervention — The intervention will consist of 4 individual telehealth parent sessions, to be completed within one month after the teen discharges from the inpatient hospital or within one month of linkage to care whatever comes first . Sessions will be 60-90 minute in length and will be offered weekly. Therapists may see parents more than once a week if needed, as long as the total number of sessions does not exceed 4.
  Arms: PI+ Inpatient Treatment as Usual
Behavioral: Treatment as usual — No parenting intervention provided beyond standard practices on the adolescent psychiatric inpatient unit.

SUMMARY:
The purpose of the present study is to conduct a pilot randomized clinical trial (RCT) of a parent coaching intervention for parents of youth hospitalized for suicidal ideation, suicide attempt(s), or non-suicidal self-injury. Parents will receive either the parent coaching intervention (which includes safety planning and behavioral parenting skills training with a clinician and assistance with linkage to follow-up care by a case manager) or treatment as usual (TAU) for the inpatient unit. The long-term goal of the research is to determine if augmenting standard inpatient treatment with additional parenting intervention improves youth treatment response on suicide-related outcomes (i.e., suicidal ideation, non-suicidal self-injury, and suicide attempts). The goal of this pilot RCT is to collect preliminary data needed for a larger RCT, including feasibility, acceptability, safety, tolerability, engagement of the presumed mechanism of change (changes in parent emotions and behaviors), and signal detection of any changes in youth suicide-related outcomes.

DETAILED DESCRIPTION:
The present study is a pilot parent coaching intervention (PI). The investigators will enroll N = 40 pairs of youth and parents enrolled in an adolescent psychiatric inpatient program. This program, called the Stanford at Mills-Peninsula Hospital (STAM), is jointly run by Stanford and Mills-Peninsula Hospital. All research procedures will be conducted by Stanford faculty and staff. Parents and youth who provide informed consent will be randomly assigned to receive the PI + standard Inpatient treatment or standard inpatient treatment only. Parents assigned to the PI + inpatient treatment will be offered 4 sessions of DBT-based parenting interventions which include safety planning, behavioral parenting interventions, and support for care linkage. Youth will participate in study assessments only and will not receive additional treatment as part of the study (i.e., they will receive treatment as usual). Study participation is optional and will not impact the family's ability to participate in the inpatient treatment. Youth will stay admitted to the inpatient program as part of standard clinical practices, regardless of whether or not they choose to participate in the study. Assessments will be conducted at baseline, 3-month follow-up, 6 month follow-up, and 12-month follow-up. Both parents will be encouraged to take part in the intervention, however; the participation of only one parent will be required. The intervention will consist of 4 individual parent sessions, to be completed within one month of youth discharge from the hospital or of care linkage whichever coms first. Sessions will be 60 to 90 minutes in length and will be offered weekly. Therapists may see parents more than once a week if needed, as long as the total number of sessions does not exceed 4. Sessions will focus on safety planning and care linkage, Parent skills building, parent conflict resolution, and parent self-care using adolescent DBT handouts.

ELIGIBILITY:
Inclusion criteria are:

* youth is currently hospitalized on the Stanford unit at Mills Peninsula Medical Center, on the Inpatient Adolescent Psychiatry Unit, for suicidal ideation and/or a suicide attempt.
* youth is between the ages of 12-18 (18 year-old youth must still be in high school and living at home with parents for the duration of the study)
* at least one parent/guardian is willing to participate in the study intervention
* youth and parent speak English well enough to complete study treatment and assessments in English

Exclusion criteria are:

• the youth or parent has a psychiatric or medical condition that would interfere with their ability to participate in study assessments and/or treatment (such as acute psychosis, neurological impairment, malnutrition due to anorexia)

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale (Posner et al., 2011) and the Suicide Attempt Self-Injury Interview (SASII; Linehan et al., 2006), Face Sheets | 3, 6, 12 months from baseline
  Structured Interviews measuring the number of suicide attempts and non-suicidal self-injury episodes
Suicide Ideation Questionnaire Jr. (Reynolds, 1988) (SIQ- Jr; Reynolds, 1988) | 3, 6, 12 months from baseline
  Self Report Measure of suicidal ideation, total score greater than 31 = clinical concern

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | 3, 6, 12 months from baseline
  Parent emotion dysregulation, higher score = greater dysregulation.
Center for Epidemiological Studies Depression Scale (CES-D, Radloff, 1977), scores range 0-60, greater than 16 = clinical concern for depressive episode | 3, 6, 12 months from baseline
  Self-report of depressive symptoms, total score of 16 or above = possible depressive episode
Caregiver Strain Questionnaire Short Form 7(CGSQ-SF7; Brannan et al., 1997) Questionnaire (CGSQ; Brannan et al., 1997) | 3, 6, 12 months from baseline
  Self-report measure of caregiver strain as a result of taking care of a child with mental health difficulties, scores range from 0-35.
Conflict Behavior Questionnaire (CBQ; Robin & Foster, 1989) | 3, 6, 12 months from baseline
  Self-report measures of family conflict, to be completed by both parents and youth, higher scores = greater conflict

CONTACTS AND LOCATIONS:
Locations (1):
- Michele Berk, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No